CLINICAL TRIAL: NCT01737671
Title: Methotrexate Infusion Into the Fourth Ventricle in Children With Malignant Fourth Ventricular Brain Tumors: A Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0823; NCI-2013-00045 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Brain Tumor; Malignant Neoplasm of Fourth Ventricle of Brain
Keywords: Brain tumor; Malignant Fourth Ventricular Brain Tumors; Ependymoma involving brain; Ependymoma involving spine; Recurrent ependymoma involving brain and/or spine; Recurrent atypical teratoid/rhabdoid tumor involving brain; Recurrent atypical teratoid/rhabdoid tumor involving spine; AT/RT; Ommaya reservoir catheter; Methotrexate; Medulloblastoma; ATRT; Atypical teratoid rhabdoid tumor; Ependymoma; Pediatric brain tumor; Intraventricular chemotherapy
MeSH Terms: conditions — Brain Neoplasms; Medulloblastoma; Rhabdoid Tumor; Ependymoma | interventions — Methotrexate; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Methotrexate Infusion (Experimental): 3 consecutive cycles of intraventricular methotrexate infusions into implanted fourth ventricle catheter/Ommaya reservoir following surgical catheter placement into fourth ventricle, each cycle is 4 consecutive daily doses of intraventricular methotrexate with minimum 2 weeks between cycles. If any serum methotrexate level is > 0.3 micromolar, then Leucovorin therapy administered (5 mg/square meter per dose) every 6 hours by vein or mouth.
  Interventions: Procedure: Ommaya Reservoir; Drug: Methotrexate; Drug: Leucovorin

INTERVENTIONS:
Procedure: Ommaya Reservoir — Surgical catheter placement into the fourth ventricle of the brain.
Drug: Methotrexate — 2 mg into fourth ventricle of the brain via the Ommaya Reservoir for 4 days. Each patient will undergo three cycles with at least two weeks between each cycle.
Drug: Leucovorin — 5 mg/square meter per dose administered every 6 hours by vein or mouth.
  Other Names: Citrovorum; Wellcovorin

SUMMARY:
The goal of this clinical research study is to learn if it is safe to receive methotrexate through the fourth ventricle of the brain in patients with brain tumors.

Methotrexate is designed to block cancer cells from dividing, which may slow or stop their growth and spread throughout the body. This may cause the cancer cells to die.

DETAILED DESCRIPTION:
Catheter Placement:

If you are eligible to take part in this study, you will have surgery to place a catheter into the ommaya reservoir. The ommaya reservoir is a catheter system that allows drugs to be administered directly to parts of the brain. In this study, the catheter will be used to collect about 1 teaspoon of cerebrospinal fluid (CSF - the fluid surrounding the brain and spinal cord) to check the status of the disease and for the infusion of methotrexate directly into the 4th ventricle of the brain, which is 1 of the 4 connected fluid-filled cavities in the brain.

If the study doctor thinks it is necessary, based on the location of the tumor, the tumor may also be removed while you are already under anesthesia just before the catheter is placed.

Study Drug Administration:

Each cycle is 4 days long and will consist of 4 daily infusions of methotrexate. You will have at least a 2 week rest period between each cycle.

Methotrexate will be infused through the ommaya reservoir catheter directly into the 4th ventricle of the brain starting at least 7 days after the catheter placement surgery. The infusion should last about 3 minutes each time.

You may also be given leucovorin, a drug used to help prevent or treat the side effects of methotrexate, by intravenous (IV) infusion through a catheter or port you have already had placed in your arm. If the study doctor thinks it is needed, this infusion will be given after each cycle to help with the possible side effects you may experience from methotrexate. The infusion should last about 5 minutes each time.

Study Visits:

Within 72 hours after catheter placement surgery:

* Any updates to your health will be recorded.
* You will have an MRI scan of the brain and spine to check the status of the disease and the flow of brain fluid.

Within seven (7) days after catheter placement surgery:

* Any updates to your health will be recorded.
* You will have a neurological exam.
* You will have a spinal tap (also called a lumbar puncture). A lumbar puncture is a procedure where fluid surrounding the spinal cord is removed by inserting a needle into the lower back. The affected area is numbed with local anesthetic during the procedure.
* You will have a neuropsychological test performed by a neuropsychologist. For this test, you will be asked questions that will test your memory and brain function. The test should take about 3 hours.

On Day 1 of each methotrexate infusion for Cycles 1-3:

* You will have a neurological exam.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* If you are able to become pregnant, you will have a urine pregnancy test.

Daily during each methotrexate infusion for Cycles 1-3:

* You will have a neurological exam.
* You will have an Ommaya reservoir tap (a catheter is placed into the Ommaya reservoir to give the methotrexate infusion).
* CSF (about 1 teaspoon) will be collected for routine tests. Blood (about 1 teaspoon each time) will be drawn to learn how much methotrexate is in your blood.

After you have completed Cycle 3:

You will have an MRI scan of the brain and spine to check the status of the disease and the flow of brain fluid.

You will have a spinal tap. You will have a neuropsychological test performed by a neuropsychologist. For this test, you will be asked questions that will test your memory and brain function. The test should take about 3 hours.

If the study doctor thinks it is in your best interest, you will continue with additional cycles of methotrexate therapy, with required tests and procedures. Your doctor may recommend additional surgery. Your doctor will discuss this with you.

Also, if the study doctor thinks it is in your best interest, methotrexate may be given together with other chemotherapy after completion of Cycle 3. If you will be receiving other chemotherapy, the study doctor will speak with you in more detail about what drugs you will receive and how you will receive them.

Length of Study:

You will receive up to 3 cycles of the methotrexate, or as long as the doctor thinks it is your best interest. You will no longer be able to receive the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after you complete the follow-up visits.

Follow-Up Visit:

3 months after the final dose of study drug:

* Any updates to your health will be recorded.
* You will have a neurological exam.
* You will have an MRI scan of the brain and spine to check the status of the disease.

This is an investigational study. Methotrexate is FDA approved and commercially available for infusion directly into brain tumors. The infusion of methotrexate into the 4th ventricle of the brain is investigational.

Up to 12 patients will be enrolled in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. There will be a two-step process of eligibility assessment: Step 1: Eligibility for catheter placement and possible surgical removal of tumor. Step 2: Eligibility for methotrexate infusion.
2. Step 1 Eligibility (Pre-Operative Eligibility) Includes: Diagnosis and Age - Patients with tumor originally located within the posterior fossa of the brain: *Patients ≤ age 21 years with recurrent medulloblastoma (PNET) involving the brain and/or spine *Patients ≤ age 21 years with recurrent ependymoma involving the brain and/or spine *Patients ≤ age 21 years with recurrent atypical teratoid/rhabdoid tumor (AT/RT) involving the brain and/or spine.
3. Step 1 Elig.: Life Expectancy - Patients must have a life expectancy of at least 12 weeks as estimated by the treating oncologist and neurosurgeon to be considered for enrollment.
4. Step 1 Elig: Central Nervous System Function - Patients may be enrolled in the study if they have an altered neurological status, such as somnolence, which is attributed to hydrocephalus and/or mass effect from the brain tumor by the treating physicians. However, after tumor resection and placement of the catheter into the fourth ventricle, the protocol will only be continued if the patient has adequate central nervous system function, defined as: patient is not severely somnolent or comatose and has adequate clinical performance status as defined in protocol section 3.2.2.1.
5. Step 2 Elig. (MTX Infusion Elig.): Clinical Performance Status - Patients must have a Lansky score of 50 or greater if ≤ 16 years of age and a Karnofsky score of 50 or greater if they are > 16 years of age to be eligible for enrollment (See Protocol Section 14.1 for Lansky Play-Performance Scale information; See Protocol Section 14.2 for Karnofsky Performance Scale information).
6. Step 2 Elig: Pregnancy - Female patients who are post-menarchal must have a negative pregnancy test to be eligible. Pregnant or lactating female patients are ineligible.
7. Step 2 Elig: Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. a. Myelosuppressive chemotherapy: Must not have received within 2 weeks of entry onto this study. b. Hematopoietic Growth Factors: At least 7 days since the completion of therapy with a growth factor. c. Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. These patients must be discussed with the study chair on a case by case basis.
8. Step 2 Elig: Bone Marrow Function - patients must have adequate bone marrow function, defined as: a. Peripheral absolute neutrophil count (ANC) ≥ 1000/µL b. Platelet count ≥ 30,000/µL (transfusion independent) c. Hemoglobin ≥ 9.0 gm/dL (may receive RBC transfusions) d. Post-op CSF flow study shows re-establishment of CSF flow.
9. All patients and/or their parents or legal guardians must sign a written informed consent.

Exclusion Criteria:

1. Patients will be excluded from this study if currently enrolled in another experimental treatment protocol.
2. Patients will be excluded from this study if they have any evidence of infection, in any site, at the time of considered enrollment.

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2012-12-27 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
Neurological Deficits After Administration of Methotrexate into the Fourth Ventricle of the Brain | 3 months
  New neurological deficit defined as new cranial neuropathy, nystagmus, change in mental status, motor deficit, or cerebellar finding (ataxia, dysmetria, dysdiadochokinesis) that is attributed by treating physicians to intraventricular methotrexate infusions.

CONTACTS AND LOCATIONS:
Overall Officials: Soumen Khatua, MD, Study Chair — M.D. Anderson Cancer Center; David Sandberg, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Children's Memorial Hermann Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org